CLINICAL TRIAL: NCT01843348
Title: 12 Month, Multi-center, Open-label, Prospective, Randomized, Parallel Group Study Investigating a Standard Regimen in de Novo Kidney Transplant Patients Versus a Certican® Based Regimen Either in Combination With Cyclosporin A or Tacrolimus
Brief Title: 12 Month Athena Study: Everolimus vs. Standard Regimen in de Novo Kidney Transplant Patients
Acronym: ATHENA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ADE44; 2011-005238-21 (EudraCT Number)
Record Dates: First submitted 2013-04-18; First posted 2013-04-30 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Kidney Transplantation; Renal Transplantation
Keywords: Transplant; Renal transplant; Rejection,allograf; Rejection; Xenograft rejection; Host vs graft disease; Kidney Transplant
MeSH Terms: conditions — Rejection, Psychology; Graft vs Host Disease | interventions — Everolimus; Tacrolimus; Cyclosporine; Mycophenolic Acid; Adrenal Cortex Hormones; Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TAC+MPA (Active Comparator)
  Interventions: Drug: Tacrolimus; Drug: Enteric Coated Mycophenolate Sodium (EC-MPS); Drug: Mycophenolate mofetil (MMF); Drug: Corticosteroids; Drug: Simulect
- TAC+Certican (Experimental)
  Interventions: Drug: Everolimus; Drug: Tacrolimus; Drug: Corticosteroids; Drug: Simulect
- CycA+Certican (Experimental)
  Interventions: Drug: Everolimus; Drug: Cyclosporin A; Drug: Corticosteroids; Drug: Simulect

INTERVENTIONS:
Drug: Everolimus
  Other Names: Certican
  Arms: CycA+Certican; TAC+Certican
Drug: Tacrolimus — Capsules: 0.5 mg, 1 mg or 5 mg. Dosing schedule: transplant to month 2: 4-8ng/ml, month 3 to month 12 3-5 ng/ml according to standard blood levels
  Arms: TAC+Certican; TAC+MPA
Drug: Cyclosporin A — Capsules: 10 mg, 25 mg, 50 mg or 100 mg. Transplantation to month 2: 75 - 125 ng/ml, month 3 to month 12: 50 - 100 ng/ml
  Arms: CycA+Certican
Drug: Enteric Coated Mycophenolate Sodium (EC-MPS) — Tablets: 180 mg or 360 mg. Dosing: duration of study 360 mg bid and no less than 360 mg daily dose
  Arms: TAC+MPA
Drug: Mycophenolate mofetil (MMF) — Capsules: 250 or 500 mg. Dosing: duration of study 500 mg bid and no less than 500 mg total daily dose
  Arms: TAC+MPA
Drug: Corticosteroids — A minimum dose of 5 mg prednisolon or equivalent
Drug: Simulect — Lyophilisate in vials with ampoules of sterile water for injection (5 mL), one vial containing 20 mg lyophilisate given intravenously on the day of transplantation and on day four post-transplantation.
  Other Names: Basiliximab

SUMMARY:
This study was designed to evaluate the renal function comparing Certican based immunosuppressive regimens with two different CNIs (Tacrolimus or Cyclosporin A) versus a standard treatment with Mycophenolic Acid and Tacrolimus in de novo renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had received a primary or secondary kidney transplant
* Patients who were willing and from whom written informed consent was obtained
* kidney allograft with a cold ischemia time (CIT) < 30 hours
* negative pregnancy test prior to study enrollment

Exclusion Criteria:

--Multi-organ recipients

* former Graft loss due to immunological reasons
* Patients who received a kidney from a non-heart beating donor
* A-B-0 incompatible transplants
* a current Panel Reactive Antibody (PRA) level of > 20%
* existing antibodies against the HLA-type of the receiving transplant
* a known hypersensitivity/contraindication to any of the immunosuppressants
* Use of other investigational drugs
* Patients with thrombocytopenia (platelets < 100,000/mm³), with an absolute neutrophil count of < 2,000/mm³ or leucopenia (leucocytes < 3,000/mm³), or hemoglobin < 8 g/dL
* significant mental illness
* history of malignancy during the last five years
* HIV positive
* uncontrolled hypercholesterolemia or hypertriglyceridemia
* drug or alcohol abuse
* pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2012-12-27 (Actual); Primary Completion 2016-03-23 (Actual); Study Completion 2016-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- France (12):
  - Novartis Investigative Site, Poitiers, France
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (15):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Tübingen

REFERENCES:
- [Derived] Philippe A, Arns W, Ditt V, Hauser IA, Thaiss F, Sommerer C, Suwelack B, Dragun D, Hillen J, Schiedel C, Elsasser A, Nashan B. Impact of everolimus plus calcineurin inhibitor on formation of non-HLA antibodies and graft outcomes in kidney transplant recipients: 12-month results from the ATHENA substudy. Front Transplant. 2023 Nov 21;2:1273890. doi: 10.3389/frtra.2023.1273890. eCollection 2023. PMID 38993854
- [Derived] Sommerer C, Suwelack B, Dragun D, Schenker P, Hauser IA, Nashan B, Thaiss F. Design and rationale of the ATHENA study--A 12-month, multicentre, prospective study evaluating the outcomes of a de novo everolimus-based regimen in combination with reduced cyclosporine or tacrolimus versus a standard regimen in kidney transplant patients: study protocol for a randomised controlled trial. Trials. 2016 Feb 17;17:92. doi: 10.1186/s13063-016-1220-9. PMID 26888217

RESULTS

PARTICIPANT FLOW:
Groups:
- TAC+MPA: Tacrolimus, Mycophenolic acid (MPA), corticosteroids and Simulect
- TAC+Certican: Tacrolimus, Certican, corticosteroids and Simulect
- CycA+Certican: Cyclosporin A, Certican, corticosteroids and Simulect
Period: Overall Study
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican
Started | 205 | 208 | 199
Safety Analysis Set (SAS) | 204 (One participant received TAC + Certican in error - analyzed with TAC + Certican arm) | 210 (Two participants received TAC + Certican in other arms in errorr - analyzed with TAC + Certican arm) | 198 (One participant received TAC + Certican in error - analyzed with TAC + Certican arm)
Full Analysis Set (FAS) | 205 (Participants in the FAS received at least one dose of study drug) | 208 (Participants in the FAS received at least one dose of study drug) | 199 (Participants in the FAS received at least one dose of study drug)
Per Protocol Set (PPS) | 147 (Participants in the FAS without major protocol deviations) | 111 (Participants in the FAS without major protocol deviations) | 80 (Participants in the FAS without major protocol deviations)
Completed | 182 | 168 | 158
Not Completed | 23 | 40 | 41
Not completed — Withdrawal by Subject | 4 | 16 | 18
Not completed — Lost to Follow-up | 5 | 4 | 2
Not completed — Death | 5 | 3 | 4
Not completed — Graft loss/retransplantation | 5 | 8 | 11
Not completed — Various reasons | 4 | 9 | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set consisted of all randomized patients who received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican | Total
Number analyzed (Participants) | 205 | 208 | 199 | 612
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (12.09) | 54.3 (13.50) | 55.1 (12.61) | 54.9 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 70 | 66 | 201
  Male | 140 | 138 | 133 | 411

OUTCOME MEASURES:

1. Primary Outcome: Glomular Filtration Rate (GFR) mL/Min Via Nankivell Method at Month 12 - Standard Regimen vs Certican Regimens
Description: To demonstrate non-inferiority in renal function assessed by glomerular filtration rate (Nankivell formula) in at least one of the Certican® treatment regimens compared to the standard regimen group at month 12 post-transplantation in renal transplant patients. Nankivell formula:
  GFR = 6.7/Scr + BW/4 - Surea/2 - 100/(height)² + C where Scr is the serum creatinine concentration expressed in mmol/L, BW the body weight in kg, Surea the serum urea in mmol/L, height in m, and the constant C is 35 for male and 25 for female patients. The eGFR is expressed in mL/min per 1.73m². If a patient was on dialysis at the time of urea or creatinine assessment, the eGFR was set to 0. Analysis set = per protocol set
Time Frame: One year post transplant
Population: Protocol analysis set comprised of participants who received at least one dose of study drug without major protocol deviaitons
Measure: Mean (Standard Deviation); unit: mL/min per 1.73m²
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican
Number analyzed (Participants) | 147 | 111 | 80
mL/min per 1.73m²
  Month 1 - Day 1 to 60 (146,111,78) | 62.62 (16.931) | 60.54 (17.310) | 59.47 (16.754)
  Month 3 - Day 61 to 136 (143,108,79) | 66.36 (16.672) | 61.21 (14.771) | 62.22 (16.196)
  Month 6 - Day 137 to 228 (142,108,76) | 68.05 (16.994) | 62.76 (16.763) | 63.17 (16.789)
  Month 9 - Day 229 to 319 (140,106,77) | 69.47 (16.251) | 64.68 (15.507) | 62.89 (14.947)
  Month12 - Day 320 to 450 (147,111, 80) | 70.41 (16.514) | 63.34 (16.986) | 61.51 (16.942)
Statistical Analysis 1: Comparison: TAC+MPA vs CycA+Certican; The trial tests the null hypotheses that the treatment difference (investigational minus reference) in mean eGFR at re-assigned visit Month 12 is lower than the non-inferiority margin (Δ) of 7 mL/min per 1.73m2 versus the alternative that the treatment difference is equal to or greater than the non-inferiority margin; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) with tx, center, donor type factors. Raw and adjusted means were presented with one-sided p-values for un-shifted and shifted hypothesis, respectively. Significance level = 2.5% (one-sided); p < 0.0001, ANOVA; Least square mean = -9.35, 95% CI 2-sided [-13.82 to -4.88]
Statistical Analysis 2: Comparison: TAC+MPA vs TAC+Certican; Test type: Non-Inferiority or Equivalence — The trial tests the null hypotheses that the treatment difference (investigational minus reference) in mean eGFR at re-assigned visit Month 12 is lower than the non-inferiority margin (Δ) of 7 mL/min per 1.73m2 versus the alternative that the treatment difference is equal to or greater than the non-inferiority margin; p = 0.0067, ANOVA — Analysis of variance (ANOVA) with tx, center, donor type factors. Raw and adjusted means were presented with one-sided p-values for un-shifted and shifted hypothesis, respectively. Significance level = 2.5% (one-sided); Least squares mean = -5.56, 95% CI 2-sided [-9.56 to -1.55]

2. Secondary Outcome: Percentage of Participants With Composite Treatment Failure Endpoints - Difference Between Groups at Month 12
Description: Combined endpoint included: biopsy proven acute rejection (BPAR) defined as a rejection which was acute and proven by biopsy, graft loss (GL) defined as: allograft was presumed to be lost on the day the patient starts dialysis and not able to be removed from dialysis or death. Patients who prematurely discontinued the study: if the patient did not suffer from an event before discontinuation and reason was not related to efficacy, the patient was assessed as having had no event, otherwise the patient was assessed as having had an event. Full analysis set (FAS)
Time Frame: Month 12 post transplant
Population: Full analysis set includes all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican | Tac+Certican - Tac+MPA - Difference Between Groups | CycA+Certican -Tac+MPA - Difference Between Groups
Number analyzed (Participants) | 205 | 208 | 199 | 413 | 404
Percentage of participants
  BPAR or graft loss or death | 9.8 | 13.0 | 24.6 | 3.2 | 14.9
  BPAR, graft loss, death, or loss of follow-up | 15.6 | 22.6 | 32.7 | 7.0 | 17.1
Statistical Analysis 1: Comparison: TAC+MPA vs TAC+Certican; TAC+Certican - TAC+MPA - difference between groups; Test type: Superiority or Other; Point estimate = 0.032, 95% CI 2-sided [-0.029 to 0.093]
Statistical Analysis 2: Comparison: TAC+MPA vs CycA+Certican; CycA+Certican -Tac+MPA - difference between groups; Test type: Superiority or Other; Point estimate = 0.149, 95% CI 2-sided [0.076 to 0.221]

3. Secondary Outcome: Glomular Filtration Rate (GFR) Via Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Method at Month 12 Post Transplant
Description: Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) method = GFR=141 x min(Scr/κ, 1)α x max(Scr/κ, 1)1.209 x 0.993Age x 1.018 [if female] x 1.159 [if black] where Scr is serum creatinine, κ is 0.7 for females and 0.9 for males, α is 0.329 for females and 0.411 for males, min indicates the minimum of Scr/κ or 1, and max indicates the maximum of Scr/κ or 1. last observation carried forward (LOCF) was used for imputation of missing values, ANCOVA model
Time Frame: Month 12 post transplant
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min per 1.73m²
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican
Number analyzed (Participants) | 181 | 166 | 158
mL/min per 1.73m² | 51.62 [48.10 to 55.14] | 44.42 [40.95 to 47.89] | 42.44 [38.89 to 45.99]

4. Secondary Outcome: Glomular Filtration Rate (GFR) mL/Min Via Cockcroft- Gault Method at Month 12 Post Transplant
Description: Cockcroft-Gault formula: For men: GFR= ((140-age) × body weight in kg)∕(72 x serum creatinine in mg∕dl)For women: GFR= (0.85×(140-age) × body weight in kg)∕(72 x serum creatinine in mg/dl), ), last observation carried forward (LOCF) was used for imputation of missing values, ANCOVA model
Time Frame: Month 12 post transplant
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min per 1.73m²
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican
Number analyzed (Participants) | 174 | 162 | 151
mL/min per 1.73m² | 60.26 [55.85 to 64.68] | 52.25 [47.88 to 56.61] | 51.30 [46.85 to 55.74]

5. Secondary Outcome: Glomular Filtration Rate (GFR) Via Modification of Diet in Renal Disease (MDRD) Method at Month 12 Post Transplant
Description: Modification of Diet in Renal Disease (MDRD) = For men: GFR = 170 x (serum creatinine -0,999) x (age-0,176) x (urea nitrogen -0,17) x (albumin0,318) For women: GFR = 170 x (serum creatinine -0,999) x (age-0,176) x (urea nitrogen -0,17) x albumin0,318) x 0.762 with urea nitrogen = urea / 2.144. last observation carried forward (LOCF) was used for imputation of missing values, ANCOVA model
Time Frame: Month 12 post transplant
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min per 1.73m²
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican
Number analyzed (Participants) | 172 | 156 | 140
mL/min per 1.73m² | 53.24 [49.62 to 56.87] | 45.72 [42.11 to 49.32] | 43.47 [39.75 to 47.20]

6. Secondary Outcome: Percentage of Participants With Treatment Failure Endpoints at Month 12
Description: Treatment failure endpoints: biopsy proven acute rejection (BPAR) defined as a rejection which was acute and proven by biopsy, graft loss (GL) defined as: allograft was presumed to be lost on the day the patient starts dialysis and not able to be removed from dialysis or death. Patients who prematurely discontinued the study: if the patient did not suffer from an event before discontinuation and reason was not related to efficacy, the patient was assessed as having had no event, otherwise the patient was assessed as having had an event. Full analysis set (FAS)
Time Frame: Month 12 post transplant
Measure: Number; unit: Percentage of participants
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican
Number analyzed (Participants) | 205 | 208 | 199
Percentage of participants
  Biopsy proven acute rejection (BPAR) | 9.3 | 12.0 | 24.6
  Treated BPAR (tBPAR) | 8.8 | 11.5 | 23.6
  Graft loss | 5.4 | 6.3 | 9.0
  Death | 4.9 | 6.3 | 6.5
Statistical Analysis 1: Comparison: TAC+MPA vs TAC+Certican; BPAR - treatment differences at Month 12; Test type: Superiority or Other; p < 0.001, Pearson's chi-square test; Odds Ratio, log = 0.028, 95% CI 2-sided [-0.032 to 0.087]

7. Secondary Outcome: Percent of Participants With Delayed Graft Function and Slow Graft Function
Description: Delayed graft function (DGF) was defined as the need for dialysis within the first 7 days post-transplantation, excluding the first post-transplantation day. Slow graft function (SGF) was defined as a serum creatinine >3.0 mg/dL at Day 5 post-transplantation. Full analysis set
Time Frame: Post transplant to month 12
Population: Full analysis set
Measure: Number; unit: Percent of participants
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican
Number analyzed (Participants) | 205 | 208 | 199
Percent of participants
  Delayed graft function (197,187,172) | 17.8 | 20.3 | 22.1
  Slow graft function (195,187,171) | 46.2 | 48.7 | 49.7

8. Secondary Outcome: Percent of Participants With Delayed Graft Function by Day
Description: Delayed graft function (DGF) was defined as the need for dialysis within the first 7 days post-transplantation, excluding the first post-transplantation day.
Time Frame: Post transplant up to day 7
Population: Full analysis set
Measure: Number; unit: Percent of participants
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican
Number analyzed (Participants) | 35 | 38 | 38
Percent of participants
  day 1 (8,7,4) | 22.9 | 18.4 | 10.5
  day 2 (2,2,2) | 5.7 | 5.3 | 5.3
  day 3 (5,1,2) | 14.3 | 2.6 | 5.3
  day 4 (4,2,4) | 11.4 | 5.3 | 10.5
  day 5 (4,5,3) | 11.4 | 13.2 | 7.9
  day 6 (1,1,2) | 2.9 | 2.6 | 5.3
  day 7 (2,4,0) | 5.7 | 10.5 | 0.0
  >7 days (9,16,21) | 25.7 | 42.1 | 55.3

9. Secondary Outcome: Percent of Participants With Viral Infections
Description: Viral infections for BKV Virus Humane Polyomavirus 1 and Cytomegalovirus
Time Frame: Post transplant to month 12
Population: Safety set
Measure: Number; unit: Percent of participants
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican
Number analyzed (Participants) | 204 | 210 | 198
Percent of participants
  Viral infections - CMVMissing | 1.0 | 0.0 | 1.0
  Viral infections - CMVAsymptomatic | 7.0 | 1.0 | 1.0
  Viral infections - CMVMild | 5.0 | 2.0 | 1.0
  Viral infections - CMVModerate | 6.0 | 1.0 | 1.0
  Viral infections - CMVSevere | 1.0 | 0.0 | 0.0
  Viral infections - BKVAsymptomatic | 10.0 | 8.0 | 5.0
  Viral infections - BKVMild | 5.0 | 7.0 | 3.0
  Viral infections - BKVModerate | 7.0 | 2.0 | 1.0
  Viral infections - BKVSevere | 0 | 0 | 0

10. Secondary Outcome: Percent of Participants With Wound Healing Complications During Study
Description: Information collected to report wound healing process which included percentage of participants with complications, fluid collections detected and occurrence of lymphoceles
Time Frame: Post transplant until individual reporting
Measure: Number; unit: Percent of participants
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican
Number analyzed (Participants) | 204 | 210 | 198
Percent of participants
  Wound healing complication | 14.3 | 19.1 | 22.2
  Fluids detected | 18.7 | 26.8 | 27.8
  Occurrence of lymphoceles | 11.8 | 18.2 | 21.8

11. Secondary Outcome: Duration of Wound Healing
Description: A wound will be considered healed if all the suture material and staples are removed and the wound is intact. Number of participants is based on all patients of the respective treatment group in the safety set, excluding patients with no answer (unknown).
Time Frame: Post transplant until individual reporting
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TAC+MPA | TAC+Certican | CycA+Certican
Number analyzed (Participants) | 28 | 34 | 38
days | 42.4 (41.13) | 54.1 (61.97) | 85.3 (62.7)

ADVERSE EVENTS:
Time Frame: Timeframe for AE
Description: AE additional description
Groups:
- Tac+MPA: Tac+MPA
- Tac+Certican: Tac+Certican
- CycA+Certican: CycA+Certican
Arm/Group | Tac+MPA | Tac+Certican | CycA+Certican
Serious Adverse Events (participants affected / at risk) | 135/204 | 161/210 | 144/198
Other Adverse Events (participants affected / at risk) | 200/204 | 205/210 | 196/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tac+MPA (N=204) | Tac+Certican (N=210) | CycA+Certican (N=198)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 0 | 1
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 5 | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphatic disorder (Blood and lymphatic system disorders) | 1 | 0 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Splenic lesion (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 2 | 3
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Cardiac flutter (Cardiac disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 2 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0 | 0
Long QT syndrome (Cardiac disorders) | 0 | 1 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Abdominal wall anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0
Parathyroid gland enlargement (Endocrine disorders) | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Anal sphincter atony (Gastrointestinal disorders) | 0 | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 2 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Drug intolerance (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Hyperthermia (General disorders) | 1 | 1 | 1
Impaired healing (General disorders) | 2 | 5 | 4
Incarcerated hernia (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 3
Oedema (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 4 | 2
Pain (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1 | 0
Chronic allograft nephropathy (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Kidney transplant rejection (Immune system disorders) | 8 | 19 | 22
Renal transplant failure (Immune system disorders) | 8 | 9 | 11
Transplant rejection (Immune system disorders) | 8 | 5 | 17
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0
BK virus infection (Infections and infestations) | 3 | 3 | 1
Bacteraemia (Infections and infestations) | 0 | 2 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 1 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 1 | 0
Cryptosporidiosis infection (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 11 | 2 | 2
Device related infection (Infections and infestations) | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 4 | 6 | 6
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 0 | 1
Epididymitis (Infections and infestations) | 0 | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 2 | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 5 | 3
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0
Graft infection (Infections and infestations) | 1 | 4 | 1
Haemophilus infection (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 0
Infected lymphocele (Infections and infestations) | 1 | 2 | 3
Infection (Infections and infestations) | 2 | 5 | 5
Influenza (Infections and infestations) | 0 | 3 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 2
Localised infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 2 | 3 | 1
Mastitis (Infections and infestations) | 0 | 0 | 1
Myocarditis infectious (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 1 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 1 | 1
Pneumonia (Infections and infestations) | 4 | 10 | 8
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1 | 1
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1
Polyomavirus-associated nephropathy (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 2
Pyelonephritis (Infections and infestations) | 10 | 9 | 8
Pyelonephritis acute (Infections and infestations) | 0 | 5 | 1
Renal abscess (Infections and infestations) | 1 | 0 | 0
Renal cyst infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Rotavirus infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 5 | 1
Septic shock (Infections and infestations) | 2 | 1 | 0
Shunt infection (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Ureteritis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 21 | 27 | 16
Urosepsis (Infections and infestations) | 9 | 6 | 7
Varicella zoster virus infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 2 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anastomotic complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 1 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 18 | 22 | 18
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 4
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 2 | 2
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 3
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Perinephric collection (Injury, poisoning and procedural complications) | 0 | 0 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 3
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 4
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Shunt aneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0
Shunt blood flow excessive (Injury, poisoning and procedural complications) | 1 | 0 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 3 | 3 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 1 | 2 | 0
Vascular graft stenosis (Injury, poisoning and procedural complications) | 2 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 3 | 3 | 4
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Anticoagulation drug level below therapeutic (Investigations) | 0 | 1 | 0
Blood creatine increased (Investigations) | 0 | 2 | 1
Blood creatinine decreased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 11 | 20 | 19
C-reactive protein increased (Investigations) | 0 | 1 | 1
Cardiac monitoring (Investigations) | 1 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0 | 0
Epstein-Barr virus antigen positive (Investigations) | 0 | 0 | 1
General physical condition abnormal (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 5 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
B-cell unclassifiable lymphoma high grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Marrow hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 0 | 2
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Device leakage (Product Issues) | 1 | 0 | 0
Device occlusion (Product Issues) | 1 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Depressive symptom (Psychiatric disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 12 | 7
Bladder pain (Renal and urinary disorders) | 0 | 1 | 0
Bladder tamponade (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 4 | 0
Micturition disorder (Renal and urinary disorders) | 1 | 0 | 0
Nephrocalcinosis (Renal and urinary disorders) | 0 | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 1 | 3
Postrenal failure (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 5 | 1
Renal artery dissection (Renal and urinary disorders) | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 4 | 2 | 2
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal haematoma (Renal and urinary disorders) | 0 | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 2 | 8 | 4
Renal infarct (Renal and urinary disorders) | 1 | 0 | 0
Renal tubular disorder (Renal and urinary disorders) | 1 | 2 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 2
Ureteral necrosis (Renal and urinary disorders) | 0 | 2 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 2 | 1
Urethral stenosis (Renal and urinary disorders) | 2 | 1 | 0
Urinary fistula (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 3 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 5 | 2
Urinoma (Renal and urinary disorders) | 1 | 1 | 2
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 2 | 3
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Renal transplant (Surgical and medical procedures) | 4 | 5 | 5
Steroid therapy (Surgical and medical procedures) | 0 | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0 | 0
Vascular anastomosis (Surgical and medical procedures) | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 3
Haematoma (Vascular disorders) | 5 | 9 | 3
Haemorrhage (Vascular disorders) | 0 | 3 | 0
Hypertension (Vascular disorders) | 0 | 2 | 1
Hypertensive crisis (Vascular disorders) | 3 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Lymphocele (Vascular disorders) | 12 | 19 | 24
Lymphoedema (Vascular disorders) | 0 | 0 | 1
Lymphorrhoea (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 1 | 0
Phlebitis deep (Vascular disorders) | 0 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 3
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tac+MPA (N=204) | Tac+Certican (N=210) | CycA+Certican (N=198)
Anaemia (Blood and lymphatic system disorders) | 44 | 53 | 58
Leukopenia (Blood and lymphatic system disorders) | 34 | 17 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 20 | 20
Tachycardia (Cardiac disorders) | 14 | 10 | 10
Abdominal pain (Gastrointestinal disorders) | 16 | 18 | 18
Abdominal pain upper (Gastrointestinal disorders) | 14 | 19 | 12
Constipation (Gastrointestinal disorders) | 71 | 69 | 81
Diarrhoea (Gastrointestinal disorders) | 19 | 17 | 6
Dyspepsia (Gastrointestinal disorders) | 14 | 17 | 9
Flatulence (Gastrointestinal disorders) | 24 | 35 | 25
Nausea (Gastrointestinal disorders) | 46 | 44 | 42
Vomiting (Gastrointestinal disorders) | 27 | 22 | 22
Impaired healing (General disorders) | 5 | 13 | 15
Oedema (General disorders) | 11 | 9 | 8
Oedema peripheral (General disorders) | 62 | 82 | 99
Kidney transplant rejection (Immune system disorders) | 8 | 9 | 14
BK virus infection (Infections and infestations) | 45 | 36 | 18
Bronchitis (Infections and infestations) | 13 | 5 | 4
Cytomegalovirus infection (Infections and infestations) | 33 | 11 | 3
Diarrhoea infectious (Infections and infestations) | 56 | 40 | 29
Nasopharyngitis (Infections and infestations) | 29 | 31 | 21
Urinary tract infection (Infections and infestations) | 81 | 74 | 72
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 28 | 36 | 43
Procedural pain (Injury, poisoning and procedural complications) | 26 | 25 | 21
Wound complication (Injury, poisoning and procedural complications) | 68 | 64 | 56
Blood creatinine increased (Investigations) | 25 | 27 | 26
Blood glucose increased (Investigations) | 6 | 15 | 8
C-reactive protein increased (Investigations) | 9 | 15 | 13
Haemoglobin decreased (Investigations) | 9 | 11 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 24 | 33 | 24
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 11 | 7
Fluid overload (Metabolism and nutrition disorders) | 7 | 7 | 13
Hypercalcaemia (Metabolism and nutrition disorders) | 16 | 16 | 13
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 16 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 20 | 25
Hyperkalaemia (Metabolism and nutrition disorders) | 65 | 53 | 58
Hyperlipidaemia (Metabolism and nutrition disorders) | 8 | 13 | 23
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 | 7 | 12
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 13 | 10
Hyperuricaemia (Metabolism and nutrition disorders) | 20 | 10 | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 20 | 27 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 33 | 37 | 41
Hypophosphataemia (Metabolism and nutrition disorders) | 23 | 36 | 30
Iron deficiency (Metabolism and nutrition disorders) | 6 | 8 | 10
Metabolic acidosis (Metabolism and nutrition disorders) | 24 | 25 | 21
Vitamin D deficiency (Metabolism and nutrition disorders) | 21 | 20 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 16 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 11 | 7
Headache (Nervous system disorders) | 15 | 25 | 15
Tremor (Nervous system disorders) | 30 | 22 | 9
Anxiety (Psychiatric disorders) | 8 | 15 | 9
Insomnia (Psychiatric disorders) | 41 | 39 | 24
Sleep disorder (Psychiatric disorders) | 22 | 21 | 22
Dysuria (Renal and urinary disorders) | 14 | 14 | 14
Haematuria (Renal and urinary disorders) | 14 | 19 | 13
Leukocyturia (Renal and urinary disorders) | 14 | 13 | 8
Nocturia (Renal and urinary disorders) | 12 | 11 | 14
Pollakiuria (Renal and urinary disorders) | 9 | 11 | 9
Proteinuria (Renal and urinary disorders) | 24 | 26 | 30
Renal impairment (Renal and urinary disorders) | 15 | 13 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 15 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 22 | 19
Acne (Skin and subcutaneous tissue disorders) | 3 | 11 | 4
Renal transplant (Surgical and medical procedures) | 8 | 9 | 17
Haematoma (Vascular disorders) | 10 | 16 | 17
Hypertension (Vascular disorders) | 52 | 62 | 57
Hypotension (Vascular disorders) | 13 | 11 | 16
Lymphocele (Vascular disorders) | 20 | 22 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trail results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigation from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., from all sites) in the clinical trial.